CLINICAL TRIAL: NCT06501885
Title: Designing an Ethnodrama Addressing PrEP Stigma Toward Young Cisgender Women in Kenya
Brief Title: PrEP (Pre-exposure Prophylaxis) Stigma and Women Ethnodrama Pre-Test Phase
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Pro00115054; R01TW012673 (NIH)
Record Dates: First submitted 2024-07-09; First posted 2024-07-15 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: HIV
Keywords: Stigma; HIV; PrEP
MeSH Terms: conditions — Social Stigma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ethnodrama Audience Members (Experimental)
  Interventions: Behavioral: Ethnodrama Intervention

INTERVENTIONS:
Behavioral: Ethnodrama Intervention — The intervention is six drama performances that are designed to transform community member beliefs about and foster support of young women's PrEP use, reduce PrEP-related enacted stigma toward young women, and reduce PrEP-related anticipated and internalized stigma among young women.

SUMMARY:
The investigators will develop and pre-test an ethnodrama intervention designed to transform community member beliefs about and foster support of young cisgender women (YCW) using PrEP.

DETAILED DESCRIPTION:
In Aim 1/Year 1, the investigators will develop the ethnodrama intervention; no data collection activities are included. In Aim 2/Year 2, the investigators will pre-test the ethnodrama intervention with invited groups of young women and members of young women's socio ecology (i.e., male partners, female peers, healthcare providers, informal community leaders, and family members).

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Young cisgender women who have taken or are taking PrEP
* Male partners of young women
* Female peers of young women
* Healthcare providers
* Informal community leaders
* Family members of young women

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Gender will be self-identified
Enrollment: 63 (Actual)
Dates: Start 2024-11-11 (Actual); Primary Completion 2025-09-03 (Actual); Study Completion 2025-09-03 (Actual)

PRIMARY OUTCOMES:
Number of participants who find the storylines and interactive components acceptable | Immediately post-intervention
  The investigators will gather feedback on the acceptability of the storylines (e.g., perceptions of whether the storylines seem real and identifiable) and interactive components (e.g., facilitated discussion).

SECONDARY OUTCOMES:
Potential effectiveness of the intervention's storylines on transforming audience members' PrEP-related perceptions as measured by a brief interviewer-administered survey using the Narrative Transportation Scale (NTS) | Immediately post-intervention
  The 12-item scale is divided into two sub-scales: engagement and personal connection. Sample items include: "I wanted to learn what happened to the women after the story ended"; "The stories in the dramas are relevant to my everyday life"; and "The stories in the drama are realistic and believable." The total score ranges from 12 to 84, where a higher score indicates greater narrative transportation.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Corneli, PhD, MPH, Principal Investigator — Duke University
Locations (1):
- Impact Research and Development, Kisumu, Kenya

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-09-15): https://cdn.clinicaltrials.gov/large-docs/85/NCT06501885/ICF_000.pdf